CLINICAL TRIAL: NCT01965132
Title: Korean College of Rheumatology Biologics and Targeted Therapy Registry
Acronym: KOBIO
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kichul Shin, Director, KOBIO registry, SMG-SNU Boramae Medical Center
Other Study IDs: KOBIO_1
Record Dates: First submitted 2013-10-11; First posted 2013-10-18 (Estimated); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
Keywords: Rheumatiod Arhthritis; Ankylosing spondylitis; Psoriatic arthritis; Biologic agents; Cohort studies; Small molecule agents
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic | interventions — Biological Products; Etanercept; Adalimumab; Infliximab; golimumab; tocilizumab; Abatacept; Rituximab; Ustekinumab; secukinumab; ixekizumab; Biosimilar Pharmaceuticals; tofacitinib; baricitinib; upadacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Biologic or targeted synthetic DMARD: Korean patients with rheumatoid arthritis, ankylosing spondylitis, and psoriatic arthritis who will initiate, restart or switch to a biologic agent (etanercept, adalimumab, infliximab, golimumab, tocilizumab, abatacept, rituximab, ustekinumab, secukinumab, ixekizumab, or biolsimilars) or a targeted synthetic DMARD
  Interventions: Drug: Biologic or targeted synthetic DMARD

INTERVENTIONS:
Drug: Biologic or targeted synthetic DMARD
  Other Names: etanercept, adalimumab, infliximab, golimumab, tocilizumab, abatacept, rituximab, ustekinumab, secukinumab, ixekizumab, or biosimilars; tofacitinib, baricitinib, upadacitinib

SUMMARY:
We established a nationwide biologics and targeted synthetic DMARDs registry (in the form of an inception cohort) to study the safety profiles in rheumatoid arthritis, ankylosing spondylitis and psoriatic arthritis patients receiving biologics or targeted synthetic DMARDs. As this registry is to observe the "real world" use of anti-rheumatic treatments under routine clinical practice, no hypothesis to prove is planned.

DETAILED DESCRIPTION:
This registry is a multi-center, prospective, observational program that will gather and analyze data on patients being treated with biologics and targeted synthetic DMARDs in Korea. In contrast to a controlled clinical trial, there is no imposed experimental intervention and solely the patients' physicians will determine the patient's treatment. Thus, the data captured and reported in this registry will reflect a "real world" approach to the treatment with biologics or targeted synthetic DMARDs. There will be no additional visit or laboratory test done outside the routine clinical practice. The selection of the agent, dosing, and treatment duration is determined by the investigator. Informed consent will be obtained from the patient prior to the collection of any data.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with RA, AS or PsA
* RA deemed by their rheumatologist to require treatment with a biologic or targeted synthetic DMARDs or a conventional DMARD(s)
* AS or PsA patients who are to initiate, restart or switch to a biologic agent or a targeted synthetic DMARD
* Patients who provide a written consent of participating in this registry (data collection and review).

Exclusion Criteria:

* RA, AS, PsA patients who are already on biologics or targeted synthetic DMARDs upon screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the following disease who will initiate, restart or switch to a biologic agent or a targeted synthetic DMARD
  1. Rheumatoid arthritis (RA)
  2. Ankylosing spondylitis (AS)
  3. Psoriatic arthritis (PsA)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2012-12-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events during the use of biologics or targeted synthetic DMARDs in Korean patients with Rheumatic diseases | up to 10 years
  Patient will be followed on a yearly basis. Adverse events based on MedDRA® during the observational period will be filled out on each follow up. Adverse events will also be assessed in the case of switching or discontinuation of biologics.

CONTACTS AND LOCATIONS:
Overall Officials: Eun Yeong Lee, MD, Principal Investigator — Seoul National University Hospital; Tae-Hwan Kim, MD, Principal Investigator — Hanyang University; Shin-Seok Lee, MD, Principal Investigator — Chonnam National University Hospital; Jaejoon Lee, MD, Principal Investigator — SAMSUNG MEDICL CENTER; Changhoon Lee, MD, Principal Investigator — Wonkwang University Hospital; Chang-Keun Lee, MD, Principal Investigator — Asan Medical Center; Hyoun-Ah Kim, MD, Principal Investigator — Ajou University School of Medicine; Sang-Il Lee, MD, Principal Investigator — Gyeongsang National University Hospital; Jung-Yoon Choe, MD, Principal Investigator — Daegu Catholic University Medical Center; Jae Hyun Jung, MD, Principal Investigator — Korea University Ansan Hospital; Mi Ryoung Seo, MD, Principal Investigator — Gachon University Gil Medical Center; Jinseok Kim, MD, Principal Investigator — Jeju National University Hospital; Mihye Kwon, MD, Principal Investigator — KONYANG UNIV. HOSPITAL; Joo-Hyun Lee, MD, Principal Investigator — Inje University Ilsan Paik Hospital; Seong Wook Kang, MD, Principal Investigator — Chungnam National University Hospital; Kwi Young Kang, MD, Principal Investigator — THE CATHOLIC UNIV. OF KOREA INCHEON ST. MARY'S HOSPITAL; Sung Won Lee, MD, Principal Investigator — Dong-A University Hospital; Young-Beom Park, MD, Principal Investigator — Severance Hospital; Hyun-Sook Kim, MD, Principal Investigator — Soonchunhyang University Hospital; Dae Hyun Yu, MD, Principal Investigator — Hanyang University; Sang-Heon Lee, MD, Principal Investigator — Konkuk University Medical Center; Young Mo Kang, MD, Principal Investigator — Kyungpook National University Hospital; Ki Won Moon, MD, Principal Investigator — KangWon National University Hospital; Seung-Jae Hong, MD, Principal Investigator — Kyunghee University Medical Center; Sang-Hyun Kim, MD, Principal Investigator — Keimyung University Dongsan Medical Center; Gwan Gyu Song, MD, Principal Investigator — Korea University Guro Hospital; Jiwon Hwang, MD, Principal Investigator — Samsung Changwon Hospital; Sung Hae Chang, MD, Principal Investigator — Soonchunhyang University Hospital; JINHYUN KIM, MD, Study Director — Chungnam National University Hospital; Joo-Hyun Lee, MD, Principal Investigator — INJE UNIVERSITY ILSAN PAIK HOSPTIAL; Wan Hee Ryu, MD, Principal Investigator — Chonbuk National University Hospital; In-Ah Choi, MD, Principal Investigator — Chungbuk National University Hospital; Hyun Ah Kim, MD, Principal Investigator — HALLYM UNIVERSITY HOSPITAL; Kichul Shin, MD, Study Chair — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government-Seoul National University Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HA, Lee E, Park SY, Lee SS, Shin K. Clinical Characteristics of Patients With Psoriatic Spondylitis Versus Those With Ankylosing Spondylitis: Features at Baseline Before Biologic Therapy. J Korean Med Sci. 2022 Aug 22;37(33):e253. doi: 10.3346/jkms.2022.37.e253. PMID 35996930
- [Derived] Kim HA, Lee E, Lee SK, Park YB, Shin K. Retention Rate and Efficacy of the Biosimilar CT-P13 Versus Reference Infliximab in Patients with Ankylosing Spondylitis: A Propensity Score-Matched Analysis from the Korean College of Rheumatology Biologics Registry. BioDrugs. 2020 Aug;34(4):529-539. doi: 10.1007/s40259-020-00432-z. PMID 32696266
- [Derived] Kim HA, Lee E, Lee SK, Park YB, Lee YN, Kang HJ, Shin K. Retention Rate and Safety of Biosimilar CT-P13 in Rheumatoid Arthritis: Data from the Korean College of Rheumatology Biologics Registry. BioDrugs. 2020 Feb;34(1):89-98. doi: 10.1007/s40259-019-00393-y. PMID 31734899
- [Derived] Kim HA, Lee E, Lee SK, Park YB, Lee YN, Kang HJ, Shin K. Retention rate and long-term safety of biosimilar CT-P13 in patients with ankylosing spondylitis: data from the Korean College of Rheumatology Biologics registry. Clin Exp Rheumatol. 2020 Mar-Apr;38(2):267-274. doi: 10.55563/clinexprheumatol/z0va6o. Epub 2019 Jul 19. PMID 31365335